CLINICAL TRIAL: NCT04882670
Title: The Impact of the COVID-19 Pandemic on Health Care and Rehabilitation Outcomes in Frail Patients With a Hip Fracture. A Retrospective Prognostic Study
Brief Title: COVID-19 Pandemic on Health Care and Rehabilitation Outcomes
Acronym: HIP COVID
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 0001531
Record Dates: First submitted 2021-02-16; First posted 2021-05-12 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Hip Fractures; Covid19
MeSH Terms: conditions — Hip Fractures; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hip fracture

SUMMARY:
Fragility fracture is easily associated with a clinical worsening of patients in terms of quality of life and disability in the medium and long term. Following this traumatic event, more than half of the patients are unable to recover pre-fracture motor skills such as the ability to walk. The impact of the COVID-19 pandemic on this type of patient has not been described and it is easy to hypothesize that, given their intrinsic frailty condition, they may have been significantly affected by changes in care pathways.

DETAILED DESCRIPTION:
The global health emergency due to the spread of COVID-19 has caused unprecedented pressure on the health systems of the various countries involved. COVID-19 has had a direct impact on the health status of people with an extremely high number of ICU admissions and deaths, but it has also led to a series of equally strong indirect consequences as described in various fields by multiple authors. In order to cope with the great health demand linked to the epidemic, hospitals had to invest human and physical resources, subtracting them from other care activities: operating theaters, surgical and non-surgical departments and the related staff normally destined for patient care were redirected and relocated to the care of COVID patients.

In the field of orthopedic surgery in the first phase of the spread of the epidemic, all non-essential interventions have been postponed and for essential interventions specific paths have been created at hospitals capable of operating even during the pandemic. This organization has led to a reduction in the overall number of hospitalized patients but the number of old patients operated for hip fracture has not decreased. From the point of view of the impact of the COVID-19 pandemic on all patients operated for hip fracture with respect to the care outcomes during the postoperative hospital stay, the available data are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with fragility hip fracture such as pertrochanteric fracture, femoral neck fracture and subtrochanteric fracture
* Age 65 or older

Exclusion Criteria:

* Patients diagnosed with a fragility hip fracture whose nursing record was not scanned at the time of the investigation
* Patients with fragility fractures of the diaphyseal and / or distal femur and acetabular fractures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: hip fracture patients who are admitted to the emergency room of an orthopedic university hospital
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of pressure ulcer | through hospitalization, an average of 9 days
  The lesions were described according to the site of onset and classified by severity categories in accordance with the guide drawn up by the National Pressure Ulcer Advisory Panel - N.P.U.A.P. (NPUAP, EPUAP, & PPPIA, 2019)

SECONDARY OUTCOMES:
Incidence of urinary infections | through hospitalization, an average of 9 days
  positive urine-culture test report
Number of accidental falls | through hospitalization, an average of 9 days
  The incidence of falls during the hospitalization
Start day for walking | through hospitalization, an average of 9 days
  The first time the patient is able to walk
Level of independence | 5 days after surgery
  ILOA scale, ranged from 0 to 50; 0 is the better level of independence and 50 the worse level of independence.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No